CLINICAL TRIAL: NCT01423721
Title: Relative Bioavailability of Bromhexine for Oral Administration of 16 mg of Bromhexine Hydrochloride Granules Compared to 16 mg of Bromhexine Hydrochloride Syrup in Healthy Male and Female Volunteers (an Open-label, Randomised, Single-dose, Replicate Design Phase I Study With Two Treatments in Four Crossover Periods)
Brief Title: Relative Bioavailability of Bromhexine Given as Granules and Syrup in Healthy Volunteers (Clinical Phase I Study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 65.129; 2011-002733-19 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-08-25; First posted 2011-08-26 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Healthy

ARMS (2):
- Bromihexine hydrochloride granules (Experimental): 16 mg granules
  Interventions: Drug: Bromihexine hydrochloride granules
- Bromihexine hydrochloride syrup (Experimental): 16 mg syrup
  Interventions: Drug: Bromihexine hydrochloride syrup

INTERVENTIONS:
Drug: Bromihexine hydrochloride syrup — syrup
  Arms: Bromihexine hydrochloride syrup
Drug: Bromihexine hydrochloride granules — granules
  Arms: Bromihexine hydrochloride granules

SUMMARY:
The objective of the current study is to investigate relative bioavailability of bromhexine hydrochloride given as granules and syrup

ELIGIBILITY:
Inclusion criteria:

- Healthy male and female volunteers

Exclusion criteria:

- Any relevant deviation from healthy conditions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
AUC0-tz (area under the plasma concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | 48 h
Cmax (maximum measured concentration of the analyte in plasma) | 48 h

SECONDARY OUTCOMES:
AUC0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to infinity) | 48 h

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 65.129.1 Boehringer Ingelheim Investigational Site, Biberach, Germany